CLINICAL TRIAL: NCT05572554
Title: The Effect of a Foot Bath on Sleep Quality in The Elderly: A Single-Blind Randomised Controlled Trial
Brief Title: The Effect of a Foot Bath on Sleep Quality in The Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Demirağ, Ph.D (Other)
Responsible Party: Sponsor-Investigator, Hatice Demirağ, Ph.D, Assistant Professor, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCS10052022
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Elderly; Sleep Quality; Complementary Therapy; Chronic Disease
Keywords: Elderly; Sleep quality; Foot bath; Complementary therapy; Chronic disease
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Disease

STUDY DESIGN:
Intervention Model Description: The sample size was calculated as 36 (18 for each group) elderly in total for the two groups (foot bath group, control group) with an effect size of 1,000 and the power of the targeted test was 0.90 (90%) in the G*Power 3.1.9.6 program with the error of α=0.05 and a reference to a previous study on the subject (14). Considering the cases such as withdrawal from the study or death during the research, each group was increased and a total of 50 elderly individuals, 25 elderly people for each group, were recruited for the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot Bath Group (Experimental): This group of elderly people were taught the foot bath practically by a researcher at the pre-study meeting and were given the "Foot Bath Information Brochure" and a "personalized water thermometer". The other researcher administered the "Elderly Information Form" and "PSQI" to all elderly people before the study using individual interviews lasting approximately 15 minutes and pen and paper method. The elderly were asked to soak their feet in the water in a marked plastic container with a depth of 10 centimeters and a temperature of 41-42°C for 20 minutes up to their ankles 50 minutes before normal sleeping hours every night for 8 weeks. In addition, the PSQI, which provides information about sleep quality, type, and severity of sleep disturbance, was applied to the elderly before the study (pretest), 4th week (interim measurement/1st measurement), and at the end of the study (8th week) for a total of 3 times during 8 weeks.
  Interventions: Other: Foot Bath Group
- Control Group (No Intervention): No application was made to the elderly in this group. Only the PSQI, which gives information about sleep quality, type, and severity of sleep disturbance, was administered to the elderly before the study (pretest), at the 4th week (interim measurement/1st measurement), and at the end of the study (8th week) for a total of 3 times for 8 weeks.

INTERVENTIONS:
Other: Foot Bath Group — The elderly were asked to soak their feet in the water in a marked plastic container with a depth of 10 centimeters and a temperature of 41-42°C for 20 minutes up to their ankles 50 minutes before normal sleeping hours every night for 8 weeks.
  Arms: Foot Bath Group

SUMMARY:
This study was carried out as a single-blind randomized controlled study to investigate the effect of a foot bath on sleep quality in the elderly.

DETAILED DESCRIPTION:
Sleep consists of psychological, physiological, and social dimensions and has an extremely significant function in meeting basic human needs. Sleep affects everyone's daily life and quality of life. One of the concepts that have been emphasized and gained importance recently is "sleep quality". Sleep quality is defined as "an individual's feeling ready and energetic for a new day after waking up". It is thought that sleep quality also has quantitative aspects such as falling asleep, sleep duration, number of awakenings at night, and subjective aspects such as restfulness or depth of sleep.

The population of elderly individuals is increasing day by day worldwide. In the changing age pyramid, the rate of elderly population was 9.7 % (8245124 people) (over 65 years of age) in 2021 and is estimated to be 11.0 % in 2025, 12.9 % in 2030, 16.3 % in 2040, 22.6 % in 2060, and 25.6% in 2080. With increasing age, changes occur in normal sleep patterns, complaints of insomnia increase, and satisfaction with sleep quality decreases. According to a literature review, sleep problems rank third among the reasons for visiting a doctor in the elderly, after digestive system problems and headache symptoms. The inability to fall asleep, waking up early in the morning, waking up frequently at night, and sleeping during the day are among the most common sleep-related problems in the elderly.

Sleep problems in the elderly can cause serious problems but are also preventable. In this sense, all health personnel, especially nurses, should apply comprehensive nursing care to minimize sleep problems and improve sleep quality in the elderly. Pharmacological treatment is generally employed in the elimination of sleep problems. However, pharmacological treatment is inadequate in eliminating sleep problems, so the elderly continuously use medication, which can cause side effects. On the other hand, the tendency toward non-pharmacological treatment has recently increased, and developments have been achieved in non-pharmacological treatment methods. It has been reported that methods such as music therapy, eye mask, complementary therapies, massage, aromatherapy, and a foot bath are used to improve the sleep quality of elderly people with sleep problems. Foot baths are reported to facilitate falling asleep by affecting body temperature. Sleep quality may improve in patients whose falling asleep process becomes easier. However, to the best of this knowledge, no study has been found in Turkey in which foot baths are used in the elderly and other populations. After all these considerations, the effect of a foot bath on sleep quality in the elderly was analyzed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years old or older,
* Being literate,
* Performing activities of daily living,
* Not having problems with the sense organs (such as eyes, ears, skin),
* Not being paraplegic/hemiplegic,
* Not working the night shift, and
* Having a mobile phone that can make video a call or having a relative with such a phone.

Exclusion Criteria:

* Refusing to participate in the research,
* Having psychological disorders,
* Using complementary therapy to sleep,
* Having enuresis,
* Being bedridden or using a wheelchair, and
* Having more than 10 years of diagnosis of diabetes or diabetes-related neuropathy.

Ages: 65 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 8 week
  PSQI is an index that questions sleep quality, type, and severity of sleep disturbance in the last month in adults. 19 questions are answered by the person himself/herself, and 5 questions are answered by the person's bedmate or people sleeping in the same room.
  The PSQI, which provides information about sleep quality, type, and severity of sleep disturbance, was applied to the elderly before the study (pretest), 4th week (interim measurement/1st measurement), and at the end of the study (8th week) for a total of 3 times during 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Demirağ, Dr.Öğr.Üyesi, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gümüşhane University, Gümüşhane, Kelki̇t, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No